CLINICAL TRIAL: NCT02765334
Title: A Pilot Feasibility Clinical Trial of Neurostyle Brain Exercise Therapy Towards Enhanced Recovery (nBETTER) for postStroke Arm Paresis
Brief Title: A Study of Neurostyle Brain Exercise Therapy Towards Enhanced Recovery (nBETTER) for Stroke
Acronym: nBETTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Institute for Infocomm Research (Other); National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2014/01164
Record Dates: First submitted 2016-04-07; First posted 2016-05-06 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2017-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Feasibility of nBETTER training (60 minutes) with conventional arm therapy (30minutes) for chronic stroke.
Oversight: Data Monitoring Committee: No

ARMS (1):
- nBETTER and Conventional Therapy (Experimental): Intervention: nBetter therapy
  Interventions: Device: nBETTER

INTERVENTIONS:
Device: nBETTER — 60 minutes of nBETTER training followed by 30 minutes of conventional therapy occupational therapy. Total of 18 sessions over 6 weeks.

SUMMARY:
A feasibility trial of Neurostyle Brain Exercise Therapy Towards Enhanced Recovery (nBETTER) system for Brain Computer Interface (BCI) neurofeedback for rehabilitation of the subacute and chronic hemiplegic upper limb aimed at improving upper limb recovery for subacute to chronic stroke patients.

DETAILED DESCRIPTION:
Stroke remains the 4th cause of death in Singapore and despite advances in neuro-medical care and rehabilitation, 40-50% of stroke survivors are left with permanent neuro-disability and a reduced quality of life. The previous 2 decades has seen exponential leaps in the development of rehabilitation technologies which enhance neuroplasticity and rehabilitation outcome. One of these potentially useful technologies is nBETTER System, was developed by Institute for Infocomm Research, Agency for Science, Technology and Research (A*STAR). nBETTER is a portable, internet-connected device that detects the imagination of movement of stroke-affected limb using a Electroencephalography (EEG)-based Brain-Computer Interface (BCI) thus delivering visually engaging feedback for directed neurofeedback aimed at improving upper limb recovery for subacute to chronic stroke patients. The pilot study aims to recruit 13 patients using a multi centre trial design to investigate nBETTER system feasibility and safety for rehabilitation of subacute to chronic stroke patients with upper limb motor impairment and to determine clinical efficacy, safety and feasibility of such a system when it is delivered with standard occupational therapy.

The investigators primary hypothesis is that nBETTER is a feasible and safe prototype in stroke survivors (> 3 months) with moderate to severe arm impairment (FMMA 10-50). The primary outcome is a gain of 15% in Fugl-Meyer motor scores at 6 weeks after 18 sessions (total of 27 hours) of supervised training by occupational therapists and bioengineers.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21-80 years with first-ever clinical stroke diagnosed on CT or MRI brain imaging.
2. Stroke duration of 3-24 months.
3. Stroke type: ischemic or haemorrhagic
4. Fugl-Meyer motor score of the upper limb range from 10-50
5. Ability to pay attention and maintain supported sitting for 1.5 hours continuously
6. Able to give own consent and understand simple instructions
7. Fulfils BCI resting brain states on initial screening.

Exclusion Criteria:

1. Recurrent clinical stroke
2. Functional status: severe aphasia or inattention, unstable medical conditions which may affect participation (e.g. unresolved sepsis, postural hypotension, end stage renal failure) or anticipated life expectancy of <1 year due to malignancy or neurodegenerative disorder)
3. Hemispatial neglect (visual or sensory) or severe visual impairment despite visual aids
4. History of epilepsy, severe depression or active psychiatric disorder
5. Skull defect or previous cranial surgery as this would affect physical fit of EEG cap interface
6. Local arm factors: severe spasticity Modified Ashworth scale >2 in any region, visual analogue scale (VAS score) >4/10, fixed joint contractures or joint replacements, patients with poor skin conditions which would contraindicate repetitive arm training.
7. TMS contraindications: females with reproductive potential not on reliable contraception; pregnancy; cardiac pacemakers; orthodontics (braces); metal implants.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-12-28 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Change in Upper extremity Fugl-Meyer motor score post training | Baseline and week 6
  As above

SECONDARY OUTCOMES:
Change in Transcranial Magnetic Stimulation Assessment (TMS) | Baseline and week 6
  As above
Change in Grip Strength | Baseline and week 6
  Grip Strength measures hand force in kgf
Change in Frenchay Arm Test of Function (FAT) | Baseline and week 6
  Frenchay Arm Test of Function (FAT) measures 5 tasks:
  * Stabilize ruler and draw line
  * Grasp and lift cylinder without dropping
  * Pick up half glass and drink
  * Replace sprung clothes peg
  * Comb hair from top down (sides and back of head)
Change in Modified Ashworth Scale score (MAS) | Baseline and week 6
  Modified Ashworth Scale score (MAS) measure spasticity of wrist and hand finger flexors on a scale from 0 to 4
Change in Visual Analogue Scale (VAS) | Baseline and week 6
  Visual Analogue Scale (VAS) measures pain on a scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Chua, MBBS, FRCP, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No